CLINICAL TRIAL: NCT05256420
Title: Effect of Kinesiotape on Postural Control in Subjects With Non-operated Anterior Cruciate Ligament (ACL) Injuries: a Randomized, Double-blind Clinical Trial
Brief Title: Effect of Kinesiotape on Postural Control in Non-operated Anterior Cruciate Ligament Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KTBALANCE080222
Record Dates: First submitted 2022-02-10; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Knee Injuries; Cruciate Ligament Rupture; Anterior Cruciate Ligament Injuries; Motor Control; Balance
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape (Experimental): Application of a kinesiotape bandage on the knee.
  Interventions: Device: Kinesiotape
- Sham Bandage (Sham Comparator): Application of a sham bandage on the knee.
  Interventions: Device: Sham Bandage

INTERVENTIONS:
Device: Kinesiotape — Application of a kinesiotape bandage on the knee.
  Arms: Kinesiotape
Device: Sham Bandage — Application of a sham bandage on the knee.
  Arms: Sham Bandage

SUMMARY:
Anterior cruciate ligament (ACL) injuries are the most common traumatic knee ligament injuries. This lesion has a devastating influence on patients' activity levels and quality of life. ACL injuries are most frequent between the ages of 15 and 45 years. Individuals who choose conservative treatment must undergo physical therapy to strengthen muscles around the knee, notably the quadriceps femoris and hamstring muscles. It had been described that in absence of surgical treatment, the knee remains unstable and vulnerable to injury having a much poorer prognosis. This study aims to analyze the effectiveness of neuromuscular taping (kinesiotape) compared to placebo in patients with non-operated anterior cruciate ligament rupture.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, diagnosed with ACL rupture (clinical and imaging) between 18 and 60 years old and not yet operated.
* Rupture isolated or combined with meniscopathy including bucket-handle.
* Partial or complete ACL rupture.

Exclusion Criteria:

* Cognitive impairment that prevents understanding of simple commands.
* Unhealed wounds in the knee complex.
* Severe skin diseases and alterations.
* Previous history of allergy to any type of bandage.
* Neurological disease with impaired balance.
* Manifest deformity of the musculoskeletal system

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-07-10 (Estimated); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
Motor Control Test (MCT) | 10 minutes
  The MCT assesses the responsiveness of the automatic motor system and recovery from unexpected perturbations of the support surface quickly and efficiently. The MCT provides latencies (time in milliseconds between the onset of translation during the MCT and the onset of the participants' response to the translational movement of the support surface). Latencies were the average of the performance of both feet.
Unilateral Stance (US). | 10 minutes
  The US balance check is a test commonly used in clinical practice to assess balance. This assessment quantifies the ability to maintain postural stability while standing on US with EO and closed. The duration of each test is 10 s. The length of each trial is 10 s. Mean center of gravity (COG) sway velocity (º/s), the ratio of the distance travelled by the COG to the time of the trial, was calculated on each leg with EO and with eyes closed (EC).
Star Excursión Balance Test (SEBT). | 10 minutes
  The SEBT is a test that provides a significant challenge to the postural control system. SEBT involves the participant maintaining a base of support with one leg while reaching maximally in different directions with the opposite leg, without compromising the base of support of the supporting leg [Gribble PA, Hertel J. Considerations for normalizing measures of the Star Excursion Balance Test. Measurement in physical education and exercise science, 2003;7(2),89-100]. This test has demonstrated high reliability of measurements, showing sensitivity in screening for functional deficits related to musculoskeletal injuries

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes